CLINICAL TRIAL: NCT07324551
Title: Microfabricated Microcatheter Advantages in Middle Meningeal Artery Embolization: an Early Experience at a Single Center
Acronym: SCIENTIA
Status: Recruiting | Type: Observational
Sponsor: Ohio State University (Other)
Collaborators: Scientia Vascular, Inc. (Unknown)
Responsible Party: Principal Investigator, Patrick Youssef, M.D, Ohio State University
Other Study IDs: 20250580
Record Dates: First submitted 2025-12-23; First posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-11

CONDITIONS: Chronic Subdural Hematoma; Hemorrhage Brain
Keywords: MMA Embolization; cSDH; Chronic Subdural Hematoma
MeSH Terms: conditions — Hematoma, Subdural, Chronic; Intracranial Hemorrhages

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: Matched pair Aristotle 14 guidewire and Plato 17 microcatheter — Participants will be randomized in 1:1 ratio to either use of study devices (matched pair Aristotle and Plato) or standard of care (surgeon combination preference) using block randomization method with a fixed block size of 4 ensuring 50% will be randomized to study devices group and 50% randomized to standard of care group.
Device: Surgeon combination preference — Surgeon will decide the on guidewire and microcatheter to use for MMA embolization

SUMMARY:
The purpose of this study is to evaluate the function of matched pair Aristotle 14 Guidewire and Plato Microcatheter in MMA embolization treatment for chronic subdural hematoma compared to surgeon's preference

DETAILED DESCRIPTION:
If you agree to take part, you will have a 50/50 chance of being assigned to one of two groups. In group 1, your procedure will use the study devices. In group 2, your procedure will use devices chosen by your surgeon. The procedure and follow up are part of standard medical care. This means that taking part in the study will not mean more time or energy compared to the usual treatment you would have.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* Patient or legally authorized representative (LAR) signs an informed consent form
* Confirmed diagnosis of subacute or chronic subdural hematoma, defined as 50% or more chronic blood
* Pre-morbid Modified Rankin Score of ≤ 3

Exclusion Criteria:

* Age < 18 years old
* Potentially dangerous anatomic variations leading to increased procedural risk or unsafe access for MMA embolization
* Unmanaged, uncontrolled bleeding disorders/blood diathesis
* Presumed septic embolus, or suspicion of microbial superinfection
* Contraindication to angiography
* CT or MRI evidence of intra-cranial tumor or mass lesion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to The Ohio State University Wexner Medical Center
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-11-03 (Actual); Primary Completion 2028-07-01 (Estimated); Study Completion 2029-07-01 (Estimated)

PRIMARY OUTCOMES:
Total Navigation/procedure time | 2 years
  Comparing between devices on both navigation and procedure time
Final Embolization Grades | 2 Years
  Comparison between device groups for final embolization grades
Incidence of AE at time of surgery | 2 Years
  Incidence of device related adverse events and incidence of procedure related adverse events
Incidence of recurrence of hemorrhage | 2 Years
  Incidence of hematoma reoccurrence/progression requiring re-intervention at 90 day follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- The Ohio State University Wexner Medical Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No